CLINICAL TRIAL: NCT00003925
Title: Phase I Study of Gemcitabine (Gemzar) and UFT/Leucovorin
Brief Title: Combination Chemotherapy In Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067112; P30CA022453 (NIH); WSU-D-1641; WSU-04-28-98-M02-FB; NCI-G99-1526
Record Dates: First submitted 1999-11-01; First posted 2003-05-02 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; Leucovorin; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium
Drug: tegafur-uracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining gemcitabine, fluorouracil-uracil and leucovorin in treating patients who have advanced cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated doses of gemcitabine, fluorouracil-uracil (UFT), and leucovorin calcium in patients with advanced refractory cancer.
* Assess the toxicity of this combination regimen in this patient population.
* Evaluate this regimen in terms of response rate, response duration, and overall survival in these patients.

OUTLINE: This is a dose escalation study of gemcitabine and fluorouracil-uracil.

Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Patients receive oral leucovorin calcium immediately followed by oral fluorouracil-uracil (UFT) three times a day on days 1-21. Courses are repeated every 28 days. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine and UFT until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy refractory to existing chemotherapy or for which no standard therapy exists
* Evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Greater than 3 months

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin greater than 8.0 mg/dL

Hepatic:

* Bilirubin less than 2.0 mg/dL
* AST less than 3.0 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No active infection requiring antibiotics
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior systemic cytotoxic chemotherapy (including fluorouracil) and recovered
* No prior gemcitabine

Endocrine therapy:

* Prior hormonal therapy allowed
* No concurrent hormonal contraception

Radiotherapy:

* At least 3 weeks since prior radiotherapy to large areas of active bone marrow and recovered

Surgery:

* Prior major surgery allowed and recovered

Other:

* No prior or concurrent antiviral nucleosides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1998-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] El-Rayes BF, Zalupski M, Shields AF, Manza SG, LoRusso P, Philip PA. A phase I study of gemcitabine and uracil-ftorfar (UFT)/leucovorin. Am J Clin Oncol. 2007 Apr;30(2):101-5. doi: 10.1097/01.coc.0000251223.98193.f4. PMID 17414457
- [Result] Philip PA, Ibrahim D, Zalupski M, Arlauskas P, Shields A. Gemcitabine and UFT plus oral calcium folinate: phase I study. Oncology (Williston Park). 1999 Jul;13(7 Suppl 3):116-9. PMID 10442378